CLINICAL TRIAL: NCT07394946
Title: Neo-Adjuvant Endocrine Therapy in Post-Menopausal Hormone Receptor Positive HER 2 Neu Negative Node Positive Early-Stage Breast Cancer Patients With One Year of Letrozole.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Care Hospital & Research Centre Foundation, Lahore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCH-001
Record Dates: First submitted 2026-01-31; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Hormone Receptor-Positive, HER2-Negative, Node Positive Breast Cancer
Keywords: Early-Stage Breast Cancer; HER2-Negative Breast Cancer; Node-Positive Breast Cancer; Hormone Receptor-Positive Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole; WW Domain-Containing Oxidoreductase

STUDY DESIGN:
Intervention Model Description: All participants will receive the same intervention - letrozole 2.5 mg orally daily for one year - and outcomes will be measured within this single group. There is no randomization, control, or comparator group, making it a single-arm study.
Masking Description: Both participants and investigators are aware that the participants are receiving letrozole.
  No placebo or comparator group is involved.
  Open-label design allows for safety monitoring and practical administration in a neoadjuvant cancer setting.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Letrozole (Experimental): Letrozole, Oral, 2.5mg daily, for 1 year
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: Letrozole — Letrozole is an oral aromatase inhibitor administered at a dose of 2.5 mg once daily for one year. It is used as neoadjuvant therapy in postmenopausal women with early-stage, hormone receptor-positive (ER+/PR+), HER2-negative, node-positive breast cancer to reduce tumor size and axillary lymph node involvement before surgery.
  Other Names: Letrozole, Oral, 2.5mg daily, for 1 year

SUMMARY:
The goal of this clinical trial is to learn whether letrozole, a hormone therapy drug, is effective in treating early-stage, hormone receptor-positive, HER2-negative breast cancer that has spread to nearby lymph nodes in postmenopausal women. The study will also evaluate the safety of taking letrozole for one year before surgery.

The main questions this study aims to answer are:

Can one year of letrozole eliminate cancer from the underarm (axillary) lymph nodes?

Can treatment with letrozole reduce the need for extensive lymph node surgery?

How safe and tolerable is long-term letrozole treatment?

This is a single-arm study, meaning all participants will receive letrozole. There is no placebo or comparison group.

Participants will:

Take letrozole 2.5 mg by mouth once daily for one year

Attend regular clinic visits for physical exams, blood tests, and imaging studies

Undergo surgery after completing treatment

Be followed for up to two years to monitor cancer recurrence and survival

DETAILED DESCRIPTION:
What is this study about?

This clinical trial is studying the use of letrozole, a hormone therapy medicine, in postmenopausal women with early-stage breast cancer that:

* Has spread to nearby lymph nodes,
* Is hormone receptor-positive (ER and/or PR positive), and
* Is HER2-negative. Letrozole is already widely used to treat hormone-positive breast cancer. In this study, it is given before surgery for a longer period than usual (one year) to see how well it works in shrinking cancer in the underarm (axillary) lymph nodes.

Why is this study being done? Many women with breast cancer that has spread to lymph nodes need axillary lymph node dissection (ALND), a surgery that removes many lymph nodes and can cause long-term side effects such as arm swelling (lymphedema), pain, and reduced arm movement.

This study aims to find out whether one year of letrozole treatment before surgery can:

* Eliminate cancer from the lymph nodes in some patients, and
* Reduce or avoid the need for extensive lymph node surgery.

Who can take part in this study?

Participants must:

* Be postmenopausal women aged 18-69 years,
* Have early-stage breast cancer (tumor size T1-T2),
* Have cancer in nearby lymph nodes (N1),
* Have hormone receptor-positive, HER2-negative breast cancer,
* Not have received prior chemotherapy or hormone therapy for this cancer. What treatment will participants receive?

All participants will receive:

* Letrozole 2.5 mg, taken once daily by mouth,
* For a total duration of one year before surgery. There is no placebo and no comparison group in this study.

What will happen during the study?

1. Screening and Baseline

   * Medical history, physical examination
   * Blood tests and breast/axillary imaging (ultrasound, mammography)
   * Confirmation of eligibility
2. Treatment Phase (1 year)

   * Daily oral letrozole
   * Regular follow-up visits for:

   Clinical assessments Imaging of lymph nodes Monitoring side effects
3. Surgery and Follow-up

   * Surgical evaluation of lymph nodes
   * Pathology testing to see if cancer remains
   * Follow-up for up to two years to monitor recurrence and survival

What are the main goals of the study? Primary goal

* To determine how many patients have no remaining cancer in the axillary lymph nodes (pathological complete response) after one year of letrozole treatment.
* To assess whether lymph node shrinkage may allow patients to avoid axillary lymph node dissection.

Secondary goals

* To measure:

  * Local or regional cancer recurrence,
  * Spread of cancer to distant organs,
  * Overall survival and disease-free survival,
  * Safety and side effects of long-term letrozole use.
* To evaluate how well ultrasound imaging predicts lymph node response to treatment.

How many participants will be included? A total of 126 patients will take part in this study.

Why is this study important?

If successful, this study may:

* Reduce the need for extensive lymph node surgery,
* Lower the risk of long-term surgical complications,
* Support a less invasive treatment approach for selected patients with hormone-positive breast cancer.

The results could help improve future treatment strategies for postmenopausal women with early-stage, node-positive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age: Patients aged 18 to 69 years.
2. Menopausal Status: All patients must be postmenopausal, confirmed by serum estradiol levels or other clinical criteria.
3. Diagnosis: Histologically confirmed infiltrating ductal carcinoma of any grade.
4. Tumor Size: Primary tumor (T) category of T1 or T2 according to AJCC 8th edition, as measured by ultrasonography (USG) and mammography.
5. Node Involvement: N1 disease documented by clinical examination and USG, with histopathology confirmed by fine-needle aspiration cytology (FNAC) or core needle biopsy.
6. Hormone Receptor Status: Patients must be estrogen receptor (ER) positive and progesterone receptor (PR) positive/negative, with HER2 status negative.

Exclusion Criteria:

1. Age: Patients aged under 18 or over 69 years.
2. Tumor Size: Patients with a primary tumor larger than T2 >5cm or with N2 disease.
3. Histological Type: Infiltrating lobular carcinoma or other non-invasive breast cancer types.
4. Prior Treatments: Previous treatment with neoadjuvant endocrine therapy (NET) or neoadjuvant chemotherapy (NACT).
5. Comorbidities: Significant comorbidities that preclude administration of anesthesia or compromise patient safety.
6. Disease Characteristics: Patients with multicentric or multifocal disease, as defined by imaging or histopathological findings.

Ages: 18 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females only
Enrollment: 126 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Extent of Axillary Nodal Pathologic Complete Response (pCR) | From baseline (pre-treatment) to the end of one-year letrozole treatment
  Proportion of postmenopausal, hormone receptor-positive (ER+/PR+), HER2-negative, node-positive breast cancer patients achieving pathological complete response (pCR) in axillary lymph nodes after one year of neoadjuvant letrozole therapy, assessed by sentinel lymph node biopsy (SLNBx).

SECONDARY OUTCOMES:
Loco-Regional Relapse Rate | Assessed at 6, 12, and 24 months post-treatment initiation
  Proportion of patients experiencing loco-regional recurrence (breast, chest wall, or axillary nodes) following one year of neoadjuvant letrozole therapy.
Distant Relapse Rate | Assessed at 6, 12, and 24 months post-treatment initiation
  Proportion of patients developing distant metastases (e.g., bone, liver, lungs) after one year of neoadjuvant letrozole therapy.
Safety and Tolerability | Monitored continuously during the 1-year treatment period, reported at 3-month intervals.
  Frequency and severity of adverse events reported by participants or observed by investigators during letrozole therapy, categorized according to CTCAE v5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Care Hospital and Research Centre Foundation, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to patient privacy and institutional data protection policies. Aggregate study results will be made publicly available through ClinicalTrials.gov and peer-reviewed publications.